CLINICAL TRIAL: NCT03052023
Title: Inguinal Hernioplasty: Comparative Study Between Laparoscopic Dual Approach, Laparoscopic Trans Abdominal Preperitoneal and Lichtenstein Procedures. A Prospective Randomized Controlled Trial
Brief Title: Comparative Study Between Lap. Dual Approach, Lap. Trans Abdominal Pre-peritoneal and Lichtenstein Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sulaiman Abdulqader Saif Alshameri, general surgeon, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHPP3
Record Dates: First submitted 2017-02-02; First posted 2017-02-14 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Inguinal Hernioplasty
Keywords: dual approach; laparoscopic hernioplasty
MeSH Terms: interventions — tetra-4-amidinophenoxypropane; Wound Healing

STUDY DESIGN:
Intervention Model Description: comparative study between three procedures of inguinal hernioplasty; open (LICHTENSTEIN), TAPP, and laparoscopic DUAL APPROACH (modified TAPP)
Who Masked: Participant, Outcomes Assessor
Masking Description: this is a randomized trial where the participants are selected randomly to each of the previous three groups , and the post operative assessment of complication and pain done by different surgical residents whom are not informed about the groups of study.
Oversight: Data Monitoring Committee: No

ARMS (3):
- group A (dual approach lap hernioplasty) (Experimental): dual approach laparoscopic inguinal hernioplasty by combination of TAPP (group B) and pneumo-dissection preperitoneal instead of sharp dissection
  Interventions: Procedure: dual approach laparoscopic inguinal hernioplasty
- group B (TAPP) (Active Comparator): trans-abdominal preperitoneal hernioplasty (TAPP) after induction of pneumoperitoneum through peritoneal approach peritoneal incision and preperitoneal dissection then mesh fixation done
  Interventions: Procedure: TAPP
- group C (Lichtenstein hernioplasty) (Active Comparator): open inguinal hernioplasty (lichtenstein) repair through inguinal incision and dissection of the sac anteriorly , excision of the sac and then mesh fixation in the posterior wall of inguinal canal
  Interventions: Procedure: (lichtenstein) repair

INTERVENTIONS:
Procedure: dual approach laparoscopic inguinal hernioplasty — after pneumoperitoneum is done preperitoneal pneumo-dissection is done and then peritoneal incision done . dissection preperitoneally and sac dissection will be easy approached
  Arms: group A (dual approach lap hernioplasty)
Procedure: TAPP — pneumoperitoneum is done and then through abdominal approach peritoneal dissection in done and sac reduction and then mesh fixation
  Arms: group B (TAPP)
Procedure: (lichtenstein) repair — inguinal incision is done and inguinal canal approach anteriorly and then sac dissection and excision then mesh fixation to posterior wall and closure the incision in layers
  Arms: group C (Lichtenstein hernioplasty)

SUMMARY:
This study designed to compare the new laparoscopic dual approach to inguinal hernia repair with trans-abdominal preperitoneal (TAPP) and lichtenstein repair (open procedure)

DETAILED DESCRIPTION:
inguinal hernioplasty is a procedures where synthetic mesh is used to strengthen the inguinal tissues sites for hernia repair different methods used which is either anterior approach (open Lichtenstein) or laparoscopic posterior approach through the abdomen (TAPP) comparing these two methods by new approach which is considered to some extent a modified TAPP by pneumo-dissection of pre-peritoneal space with abdominal approach by lap. repair

ELIGIBILITY:
Inclusion Criteria:

* Adult male patient (older than 18y).
* Not complicated.
* No previous lower abdominal incisions (lower abdominal midline and lower paramedian incision in the same side of hernia).
* No contraindication for general anesthesia.
* Not recurrent.

Exclusion Criteria:

* any one not in fulfill inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
operative time | from the inflation of the abdomen till deflation and port closure ---for lichtenstein from skin incision to skin closure.
  operative time will be measured in minutes for each procedure.and comparing three groups ( dual approach , TAPP and Lichtenstein ) in operative time which determined as follow:
  * from the inflation of the abdomen till deflation and port closure
  * for Lichtenstein from skin incision to skin closure

SECONDARY OUTCOMES:
intraoperative injuries | intra operative
  abdominal visceral injuries cord structure injuries
intra operative bleeding | intraoperative
  mild bleeding and oozing controlled by cautery bleeding from inferior epigastric artery or testicular artery major vascular injury
post operative pain | immediately post operative and 6 ,12, 24 hours and two weeks post operative
  pain measured by visual analog scale from 0 no pain to 10 the worst pain ever.
post operative wound complication | 2 weeks post operative ,3 ,6 and 12 months postoperative
  wound seroma , hematoma either small with conservative treatment and large need intervention wound infection either superficial skin and S.C. or mesh infection
post operative chronic pain | follow up at 3 months , 6 months and one year for pain assessment by VAS
  post operative paraesthesia , bricking pain, dull-aching pain. measured by visual analog scale (VAS) from 0 no pain to 10 the worst pain ever
recurrence | 3 months, 6 months and one year
  post operative inguinal swelling confirmed clinically as a recurrent hernia

CONTACTS AND LOCATIONS:
Overall Officials: mostafa A. hamad, professor, Principal Investigator — Assiut university hospital faculty of medicine
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nasr MM. Early results of dual approach hernioplasty (DAH): an innovative laparoscopic inguinal hernioplasty technique. Surg Endosc. 2016 Mar;30(3):1113-8. doi: 10.1007/s00464-015-4308-5. Epub 2015 Jun 23. PMID 26099622